CLINICAL TRIAL: NCT02159768
Title: Visualization of the Larynx With the Airtraq Laryngoscope and Image Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/00376
Record Dates: First submitted 2014-06-09; First posted 2014-06-10 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Anaesthesia
Keywords: tracheal intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Airtraq visualization (Experimental): Larynx visualization with Airtraq and attached handphone
  Interventions: Device: Airtraq visualization

INTERVENTIONS:
Device: Airtraq visualization — Larynx visualization with Airtraq and attached handphone
  Other Names: Airtraq Avant

SUMMARY:
The Airtraq is a battery powered single use optical laryngoscope with a channel to hold and guide the tracheal tube into the trachea. It enables tracheal intubation in patients with normal and difficult airways, by enabling laryngoscopy without neck movement. As a single use device, it is cost effective to have these placed in emergency equipment kits, and for use by emergency and military personnel.

However, it does have several limitations. The Airtraq requires the user to place his/her eye to the eyepiece in order to see the advancement of the laryngoscope and the tracheal tube, which may be difficult if the patient is on the ground or in emergency scenarios. Only the user can see through the eyepiece and any assistants are unable to view the larynx, this makes it difficult for assistants to help the operator.

Many handphones now incorporate high quality cameras. In this study, we will evaluate the effectiveness of using the iPhone to aid laryngoscopy with the Airtraq optical laryngoscope during laryngoscopy and intubation in 30 patients presenting for elective surgery under general anaesthesia. We have manufactured an attachment that fits over the eyepiece of the Airtraq, to hold an iPhone to the eyepiece. This will enable to operator and assistants to simultaneously view the insertion of the Airtraq, view the larynx and view the passage of the tracheal tube into the trachea.

DETAILED DESCRIPTION:
This study is a single-cohort study design. 30 patients undergoing elective surgery under general anaesthesia will be recruited. They will have endotracheal intubation done with the Airtraq optical laryngoscope and handphone camera assisted visualization.

The Airtraq optical laryngoscope fitted with the attachment holding the camera handphone will be prepared and loaded with an appropriately sized endotracheal tube. A standard general anaesthesia technique will be used. This will include standard monitoring including pulse oximetry, non-invasive blood pressure, ECG and capnography, all started before induction of anaesthesia. Anaesthesia will be induced with proprofol and fentanyl, and muscle relaxation with atracurium.

The airway management procedure will start after induction of anaesthesia and muscle relaxation. The Airtraq optical laryngoscope will be used. The Airtraq is fit with an attachment to hold the camera handphone, and loaded with an endotracheal tube. The Airtraq will be inserted and manipulated until the best view of the patient's laryngeal opening can be seen on the camera handphone screen. The endotracheal tube will then be placed in the patient's trachea and the cuff inflated. Successful intubation will be confirmed by 3-point auscultation and presence of end-tidal carbon dioxide tracing.

ELIGIBILITY:
Inclusion Criteria:

Adult patients requiring general anaesthesia for elective surgery and who require tracheal intubation as part of the anaesthesia technique.

American Society of Anesthesiologists Class I to III physiological status.

Exclusion Criteria:

Children Pregnant patients Patients who have not fasted for at least 6 hours pre surgery Patients at risk of regurgitation and aspiration

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene H Liu, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 16 July 2014 to 27 July 2015, in hospital ward, before surgery and anesthesia.
Period: Overall Study
Arm/Group | Airtraq Visualization
Started | 30 (Started 16 July 2014)
Completed | 30 (Completed 27 July 2015)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Airtraq Visualization
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Region of Enrollment [Number; unit: participants]
  Singapore | 30

OUTCOME MEASURES:

1. Primary Outcome: Visualization of Larynx With the Airtraq Laryngoscope and Handphone
Description: The efficacy of viewing the larynx via the handphone attached to the Airtraq laryngoscope will be assessed.
Time Frame: Intra operative
Population: Study participants in whom the Airtraq handphone visualization system was studied
Measure: Number; unit: participants
Arm/Group | Airtraq Visualization
Number analyzed (Participants) | 30
participants | 30

2. Secondary Outcome: Transmission of Airtraq View of Larynx
Description: The view of the larynx will be captured by the handphone attached to the Airtraq layryngoscope, and then transmitted to a second investigator.
Time Frame: Intra operative measurement, time frame within 5 minutes
Population: The larynx could be visualized in all 30 patients using the handphone attached to the Airtraq. The images of the larynx could be transmitted to a remote assistant in all 30 patients.
Measure: Number; unit: participants
Arm/Group | Airtraq Visualization
Number analyzed (Participants) | 30
participants | 30

ADVERSE EVENTS:
Time Frame: 1 year 3 months.
Arm/Group | Airtraq Visualization
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No